CLINICAL TRIAL: NCT02019940
Title: An Investigation of the Effects of Riluzole in Patients With Post-Traumatic Stress Disorder (PTSD)
Brief Title: A Pilot Study Of Riluzole In Patients With Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for PTSD (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1308012549
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Riluzole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Riluzole (Experimental): Riluzole 50 mg orally twice per day
  Interventions: Drug: Riluzole

INTERVENTIONS:
Drug: Riluzole

SUMMARY:
This open label study will evaluate the safety and efficacy of riluzole in patients with PTSD. Patients will receive riluzole 50mg twice per day orally for 12 weeks as outpatient, with a one month follow up at week 16.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18-75 years;
* Able to provide written informed consent;
* Current Post Traumatic Stress Disorder, as determined by the Clinician Administered Scale for PTSD, or the presence of sub-threshold PTSD. Individuals with sub-threshold PTSD will be included at the discretion of the PI;
* Clinician Administered PTSD Scale (CAPS) score of 23 or higher;
* Be able to understand and speak English.
* Subjects taking FDA-approved antidepressant medications may enter the study if they have been on a stable dose for at least 4 weeks prior to starting the study drug.

Exclusion Criteria:

* Breastfeeding women and pregnant women, or women of child bearing potential who are not using a medically accepted means of contraception (to include oral, injectable, or implant birth control, condom, diaphragm with spermicide, intrauterine device, tubal ligation, abstinence, or partner with vasectomy);
* Current, ongoing serious suicidal risk as assessed by evaluating investigator or by scoring 5 or more on the item-10 of the MADRS.
* Unstable medical illness as determined by the investigator;
* Patients with schizophrenia or schizoaffective disorders (current or past);
* Substance use disorder during the 3 months prior to screening; except for Cannabis and Alcohol use Disorders.
* Clinical evidence of untreated hypothyroidism;
* Patients with any evidence of clinically significant liver abnormalities, or any liver transaminase level > 1.5 x ULN at initial screening, or > 5 x ULN during treatment;
* Axis II personality disorders that are the primary purpose of treatment, or would interfere with a patient's safety or compliance, as determined by the investigator during open-ended psychiatric interview;
* Patients currently being treated for a respiratory disorder (including asthma or COPD);
* For participants over the age of 60, evidence of dementia as determined by the St. Luis University Mental Status Exam (SLUMS; participants with total scores less than or equal to 20 will be excluded and referred to their Primary Care Physician for follow-up/dementia evaluation); Structured psychotherapy focused on treatment of PTSD is exclusionary unless the subject has had at least 8 weeks of treatment prior to starting the study medication;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Abdallah, MD, Principal Investigator — National Center for PTSD / Yale University
Locations (1):
- Clinical Neuroscience Division, National Center for PTSD, West Haven, Connecticut, United States

REFERENCES:
- See also: National Center for PTSD — http://www.ptsd.va.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Riluzole Open Label: Subjects diagnosed with PTSD will receive riluzole, 50 mg taken orally twice daily (BID) for 12 weeks
Period: Overall Study
Arm/Group | Riluzole Open Label
Started | 18
Completed | 8
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: 18 participants started the study and 9 participants were randomized into the single arm of the study. However, only 8 participants completed the treatment. Since there was some treatment data collected on the 9th participant, he/she was included in the analysis.
Arm/Group | Riluzole Open Label
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Indication of whether a participant is male or female
  Participants
    Female | 2
    Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician Administered PTSD Scale (CAPS)
Description: The CAPS is a standardized clinician-rated instrument to assess the presence and severity of PTSD symptoms. The scores range from 0 (minimum) to 80 (mazimum). Higher scores reflect worse symptoms.
Time Frame: Change from baseline to 12 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole Open Label
Number analyzed (Participants) | 9
units on a scale | -20.67 (21.16)

2. Secondary Outcome: Post-Traumatic Stress Disorder Checklist (PCL)
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Clinical Global Impressions Scale
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Quick Inventory of Depressive Symptoms - Self-Report (QIDS-SR)
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: The reporting of the adverse events reflects that one participant could have experienced more than one adverse event. For example, one participant experienced both dry mouth and lightheadedness. Similarly, three participants could have experienced chest pain. Thus, it may seem like the number of participants that experienced various adverse events does not match up to the number of participants in the participant flow. We analyzed 9 participants total and recorded their AEs in this section.
Arm/Group | Riluzole Open Label
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 7/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riluzole Open Label (N=9)
Abdominal Pain (General disorders) | 1
Dry mouth (General disorders) | 2
Altered Taste Sensation (General disorders) | 1
Light headedness (General disorders) | 2
Headache (General disorders) | 2
Rhinitis, congestion, sinus pressure, postnasal drip (General disorders) | 1
bruxism (General disorders) | 1
fatigue (General disorders) | 3
chest pain (General disorders) | 3
dry cough (General disorders) | 1
urinary urgency (General disorders) | 1
edema (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT02019940/Prot_SAP_000.pdf